CLINICAL TRIAL: NCT01504035
Title: Effectiveness of the Addition of Lidocaine to a Hemostatic, Bioresorbable Putty in the Treatment of Iliac Crest Donor Site Pain
Brief Title: Analgetic Effectiveness of a Lidocaine Loaded Hemostatic, Bioresorbable Putty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Orthocon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORG 001
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Pain
Keywords: Donor site pain; Iliac crest; Bone graft; Hemostatic putty; lidocaine; Donor site pain following harvest of iliac crest bone grafts
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemostatic putty plus Lidocaine (Orthostat-L) (Experimental)
  Interventions: Device: Orthostat-L
- Hemostatic putty (Orthostat) (Active Comparator)
  Interventions: Device: Orthostat

INTERVENTIONS:
Device: Orthostat-L — Application of nx2g Lidocaine loaded hemostatic putty, i.e. Orthostat-L at the iliac crest bone graft harvest site
  Other Names: Xybrex
  Arms: Hemostatic putty plus Lidocaine (Orthostat-L)
Device: Orthostat — Application of nx2g hemostatic putty, i.e. Orthostat at the iliac crest bone graft harvest site
  Other Names: Hemabsorb
  Arms: Hemostatic putty (Orthostat)

SUMMARY:
The goal of this study was to test the efficacy of local analgesic (lidocaine) loaded hemostatic putty in reducing donor site pain following the harvest of pelvic bone grafts. In 14 patients undergoing harvest of a pelvic bone graft during foot surgery, the bone defect at the pelvis was either filled with a lidocaine loaded hemostatic putty (Orthostat-L) or the same putty without lidocaine (Orthostat, currently marketed as Hemabsorb). Postoperatively, foot pain was eliminated with a peripheral nerve block, while pelvis pain was quantified with two commonly used pain rating scales (VAS and Wong Baker). Blood samples were collected at regular time intervals to measure lidocaine levels. Patients which received the lidocaine loaded putty experienced significantly less pain during the first 12 hours after surgery as compared to those patients who received the lidocaine deficient putty. Blood lidocaine levels always stayed below the toxic threshold.

DETAILED DESCRIPTION:
The harvest of iliac crest bone grafts (ICBG) is associated with relevant donor site pain, but may be lowered by the local application of a biodegradable, hemostatic putty loaded with Lidocaine (=Orthostat-L ™) for sustained local analgesic release. The primary goal of this double-blind controlled trial was to assess the efficacy of the addition of Lidocaine to a hemostatic putty in reducing donor site pain following ICBG in foot and ankle procedures.

In 14 patients undergoing ICBG harvest during a foot and ankle procedure, the bone defect at the iliac crest was either filled with Orthostat-L™ (n=7) or with the same hemostatic putty without Lidocaine (Orthostat ™, n=7; currently marketed as HemasorbTM). Postoperatively, donor site pain was managed by patient controlled morphine delivery while surgical site pain was eliminated by a peripheral nerve block. During the first 72 postoperative hours, donor site pain was quantified every 4 hours using a Visual Analog Scale (VAS) and the Wong Baker FACES pain rating scale. In addition, cumulated morphine doses required by the patients and serum Lidocaine levels were registered. Pain scores were plotted over time to calculate the area under the curve (AUC) as a representative of the overall pain experienced within specific time points.

There were no significant differences in bone graft size, putty amount and cumulated morphine use between the two groups. Orthostat-L™ provided a significant overall harvest site pain reduction over the first 12 hours postoperatively as evidenced by a significant decrease of the AUC in both VAS and Wong Baker FACES pain score plots (p=0.0366 and p = 0.0024, respectively). After 12 hours, pain scores rapidly returned to baseline levels in both groups. Serum Lidocaine consistently remained below the level of toxicity of 6mg/l.

In conclusion, the addition of Lidocaine to a hemostatic putty offers a significant ICBG harvest site pain reduction over the first 12 postoperative hours and appears to be safe in clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for a foot and ankle procedure that requires harvest of an iliac crest bone graft
* Written informed consent
* No child bearing potential

Exclusion Criteria:

* History of iliac crest bone graft removal
* Liver failure
* Heart failure
* Mental condition impeding cooperation in the study ( e.g. dementia)

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pelvic Donor Site Pain quantified by the VAS and Wong Baker Pain Rating Scale | 72 hours after putty administration
  Pain scores were plotted over time to either quantify pain at specific time points or to calculate the area under the curve in between two time points as a representative of the overall pain experienced in a specific time intervall.

CONTACTS AND LOCATIONS:
Overall Officials: Valderrabano Victor, MD PhD, Principal Investigator — Orthopedic Department, University Hospital Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Wang CF, Djalali AG, Gandhi A, Knaack D, De Girolami U, Strichartz G, Gerner P. An absorbable local anesthetic matrix provides several days of functional sciatic nerve blockade. Anesth Analg. 2009 Mar;108(3):1027-33. doi: 10.1213/ane.0b013e318193596a. PMID 19224820
- [Background] Wang CF, Pancaro C, Gerner P, Strichartz G. Prolonged suppression of postincisional pain by a slow-release formulation of lidocaine. Anesthesiology. 2011 Jan;114(1):135-49. doi: 10.1097/ALN.0b013e3182001996. PMID 21169797
- [Derived] Muller MA, Mehrkens A, Zurcher R, Vavken P, Valderrabano V. Effectiveness of the addition of Lidocaine to a hemostatic, bioresorbable putty in the treatment of iliac crest donor site pain. BMC Musculoskelet Disord. 2014 Dec 8;15:415. doi: 10.1186/1471-2474-15-415. PMID 25482244